CLINICAL TRIAL: NCT00715026
Title: Multicenter Post Approval Study of the Trilogy AB(R) Acetabular System
Brief Title: Trilogy AB Acetabular Hip System Post Approval Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor business decision unrelated to clinical performance.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-300; 06-300, Revised 3-1-2010 (Other: Zimmer - revision date)
Record Dates: First submitted 2008-07-08; First posted 2008-07-15 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Osteoarthritis; Avascular Necrosis; Congenital Hip Dysplasia; Traumatic Arthritis
Keywords: Arthritis; Total Hip; Ceramic; Hip Replacement; Total Hip Arthroplasty (THA); Joint Disease
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital; Arthritis; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trilogy AB Acetabular Hip Implant System (Other): Post Approval Study of Device.
  Interventions: Device: Trilogy AB Acetabular Hip Implant System

INTERVENTIONS:
Device: Trilogy AB Acetabular Hip Implant System — Total hip replacement with ceramic on ceramic treatment surfaces.

SUMMARY:
This is a post-approval study with prospective enrollment in the United States and a retrospective enrollment outside the United States to obtain functional, quality of life and radiographic data, which will facilitate assessment of the clinical performance of the Zimmer Trilogy AB Acetabular Hip System.

DETAILED DESCRIPTION:
To obtain functional, quality of life and radiographic data to evaluate the clinical performance of the Zimmer Trilogy AB Acetabular Hip System in primary total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese patients
* The patient is a good candidate for a primary hip arthroplasty using the Zimmer Trilogy AB Acetabular Hip System.
* Patient is willing and able to give informed consent to participate in the follow-up program.
* Patient is suitable for surgery and able to participate in the follow-up program.

Exclusion Criteria:

* Skeletally immature
* Rheumatoid arthritis
* Osteoradionecrosis
* Infection
* Nerve or muscle disease that may have a negative affect on gait or weight bearing
* Loss of abductor musculature in the affected limb
* Poor bone stock
* Poor skin coverage around the hip joint
* Rapid disease progression as obvious by joint destruction or bone absorption seen on x-ray
* Previous total or cemented hemi-arthroplasty of the affected hip
* Previous pinning or plating of the affected hip
* Patients with heavy labor jobs or extreme activity levels
* Patients who participate in sports activities or require deep flexion
* Patients who are obese
* Patients who have other disabilities
* Patients who are unwilling or unable to give consent, or to comply with the protocol and follow-up program.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Schrock, MD, Principal Investigator — Schrock Orthopedic Research; Gwo-Chin Lee, MD, Principal Investigator — University of Pennsylvania/Penn Presbyterian Hospital
Locations (2):
- United States (2):
  - Shrock Orthopedic Research, Fort Lauderdale, Florida
  - University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Trilogy AB Acetabular Hip Implant System: Post Approval Study of Device.
  Trilogy AB Acetabular Hip Implant System : Total hip replacement with ceramic on ceramic treatment surfaces.
Period: Overall Study
Arm/Group | Trilogy AB Acetabular Hip Implant System
Started | 31 (30 unilateral subjects and 1 bilateral)
Subjects That Received Surgery | 25 (24 unilateral subjects and 1 bilateral)
Completed | 21 (20 unilateral subjects and 1 bilateral)
Not Completed | 10
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 1
Not completed — Surgery done on non-study consented hip | 1

BASELINE CHARACTERISTICS:
Arm/Group | Trilogy AB Acetabular Hip Implant System
Number analyzed (Participants) | 25
Age, Continuous [Median (Standard Deviation); unit: Years] | 58 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score
Description: The Harris Hip Score was developed to assess hip disabilities and methods of treatment and has been in use for decades. It evaluates patients on the basis of pain, function, absence of deformity and range of motion. The Harris Hip Score could range from 0 to 100. Scores less then 70 are poor, scores 70 to 79 are fair, scores 80 to 89 are good, and scores 90 to 100 are excellent.
Time Frame: Pre-op, 3 Month Post-Op and Annual Post-Op visits through 5 Years
Population: Data was received on 24 subjects/25 hips at preop, on 17 subjects/18 hips at 3 months, and on 4 subjects at 1 year prior to the early termination of the study. Each hip, whether unilateral or bilateral, was counted separately. Early study termination was done due to voluntary removal of the device from the US market.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trilogy AB Acetabular Hip Implant System
Number analyzed (Participants) | 24
units on a scale
  Preop Harris Hip Scores | 52.7 (11.6)
  3 Months Harris Hip Score | 68.2 (16.11)
  1 Year Harris Hip Scores | 70 (19.54)

2. Secondary Outcome: Continued Assessment of Implant Survivorship and Incidences of Adverse Events.
Description: A total of 37 Adverse Events were reported. There have been no UADEs reported in this study population. At the time of site closure all AEs were resolved or tolerated. Implant survivorship not reportable due to early study termination.
Time Frame: At all follow-up visits through 5 Years and postcard follow-up 6 - 10 Years
Measure: Number; unit: adverse events
Arm/Group | Trilogy AB Acetabular Hip Implant System
Number analyzed (Participants) | 25
adverse events
  SAEs - Not device related | 11
  AEs - Not device related | 21
  AEs - Definitely device related | 3
  AEs - Uncertain relation to device | 2

ADVERSE EVENTS:
Description: Of the Serious Adverse Events, all were not related to the device. Of the other Adverse Events 3 were related to device and 2 were uncertain in relation.
Arm/Group | Trilogy AB Acetabular Hip Implant System
Serious Adverse Events (participants affected / at risk) | 6/25
Other Adverse Events (participants affected / at risk) | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilogy AB Acetabular Hip Implant System (N=25)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Other/General (General disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Contralateral Hip Replacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
GI Bleed (Gastrointestinal disorders) | 1 (1)
Respiratory Failure/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pre-Renal Azotemia (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trilogy AB Acetabular Hip Implant System (N=25)
Rash/Skin Lesions (Skin and subcutaneous tissue disorders) | 1 (2)
Infection/Fever/Drainage (Infections and infestations) | 2 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Thigh/Hip/Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — Both instances of Thigh/Hip/Groin Pain were uncertain in the relation to the device.
Femur Fracture (Musculoskeletal and connective tissue disorders) | 3 (3) — All 3 femur fractures were definitely related to the device
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oxygen Desaturation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Electrolyte Imbalance (General disorders) | 2 (2)
Alcohol Abuse/Withdrawal (General disorders) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
A business decision unrelated to device performance led to the early termination of the study and withdrawal of the study device(s) from the US market. Early termination of the study limits the usefulness of the available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No